CLINICAL TRIAL: NCT02141568
Title: Effectiveness and Cost-Effectiveness Analysis of Mind-Body Interventions in a Multi-Disciplinary Clinic for Frequent Attendees Suffering From Medically Unexplained Symptoms (MUS)
Brief Title: Effectiveness of Mind-Body Interventions for Frequent Attendees Suffering From Medically Unexplained Symptoms (MUS)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low patient compliance and dropout during the period defined for the study
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-016312-CTIL; SCRC12014 (Other: Soroka Clinical Research Center (SCRC))
Record Dates: First submitted 2014-05-15; First posted 2014-05-19 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-03

CONDITIONS: Neurasthenia; Chronic Pain; Chronic Headache
Keywords: Cost-effective; Unexplained Medical Symptoms; Frequent Attenders
MeSH Terms: conditions — Neurasthenia; Chronic Pain; Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group for Prospective Study (Experimental): Intervention: Medical and psychological treatment at the Soroka UMC "functional neurology" outpatient clinic. Treatment will be conducted by a multidisciplinary staff. Patients will undergo an initial meeting with a neurologist and afterwards will be directed to other members of the team (psychologist, physical therapist) on a case by case basis.
  Interventions: Other: Medical and Psychological treatment
- No Intervention (No Intervention): Patient records will be analyzed via Clalit Health Service electronic records. No additional intervention will occur

INTERVENTIONS:
Other: Medical and Psychological treatment — Medical and psychological treatment by the staff of the "functional neurology" clinic at Soroka UMC. This treatment will include an initial visit to the staff neurologist and further multidisciplinary treatment as per his decision (the team includes a psychologist and a physical therapist).
  Arms: Intervention Group for Prospective Study

SUMMARY:
The purpose of this study is to check the medical efficacy and economic benefits of multidisciplinary care in patients with unexplained medical complaints and consume medical services frequently.

DETAILED DESCRIPTION:
Background:

Somatic or "medically unexplained" symptoms and syndromes are common and are seen by physicians across almost every medical specialty. In many instances, these phenomena can cause a great deal of pain and frustration, restrict function and reduce patients' quality of life. Despite their frequency and severity, medical personnel often experience a great deal of difficulty in coping with such complaints and patients may be shuttled from specialist to specialist, often with little or no symptomatic relief and at a great deal of expense to the medical system. Many researchers now believe that these seemingly unrelated and "unexplained" conditions in fact share common psycho-physiological mechanisms, such as being catalyzed as a result of trauma or excessive stress, being mediated by the limbic system and affecting inhibitory sensory pathways.

Purpose of the study:

Testing the efficacy and cost-efficiency of a holistic multidisciplinary treatment methodology for medically unexplained symptoms (MUS).

Stages of the Study:

The study wil lbe conducted via two arms:

1. A reterospective study of patients attending the Functional Neurology clinic a Soroka UMC between the years 2014-2018 in which patient records will be obtained via the regional offices of Clalit Health Services and analyzed in order to learn the effects of mind-body therapies on health care utilization.
2. A prospective study of new patients arriving at the "functional neurology" clinic at Soroka UMC. Members of the second arm will be asked if they would be willing to participate in the study by their neurologist. Participants who have agreed to join the study will fill out Self-report measures at the beginning of their treatment, at the end of treatment (3 months) and 6 months after the start of treatment and 12 months after the start of treatment.

Expected Results

1. A decrease in expense rates and use of medical services
2. An increase in patient satisfaction
3. An increase in patient-reported health and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* Age 18 or higher
* Treated at the Functional Neurology clinic at Soroka UMC

Exclusion Criteria:

* patients with chronic illness such as cancer, dialysis patients, or any other severe identified illness
* patients who do not speak Hebrew
* bedridden patients
* Schizophrenia, dementia and other severe mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Health Related Quality of Life | 6 months
  Changes in the Short Form 36 Health Survey (SF-36)

SECONDARY OUTCOMES:
Cost-effectiveness | 12 months
  Total cost associated with healthcare due to intervention
Anxiety | 6 months
  Changes in the State-Trait Anxiety Inventory (STAI)
Depression | 6 months
  Changes in the Patient Health Questionnaire 9 (PHQ-9)
Catastrophization | 6 months
  Changes in the Pain Catastrophization Scale (PCS)
Locus of Control | 6 months
  Changes in the Health Locus of Control Survey (H-LOC)
Existence of Symptoms | 6 months
  Changes in the Patient Health Questionnaire 15 (PHQ-15)
Pain Symptoms and Functioning | 6 months
  Changes in the Short Form Treatment Outcomes in Pain Survey (S-TOPS)
Patient Satisfaction with Medical Care | 6 months
  Changes in the Low Threshold Experience Survey (LTES)

CONTACTS AND LOCATIONS:
Overall Officials: Yacov Ezra, MD, Principal Investigator — Soroka University Medical Center
Locations (1):
- Soroka University Medical Center, Beersheba, Israel